CLINICAL TRIAL: NCT05898282
Title: Prevalence and Associated Factors of Anesthetic Drug Administration Error Among Anesthetists Working in Teaching and Referral Hospitals of Ethiopia, a Web Based Crossectional Survey, 2022.
Brief Title: Prevalence and Associated Factors of Anesthetic Drug Administration Error, a Web Based Crossectional Survey, 2022.
Status: Completed | Type: Observational
Sponsor: DebreTabor University (Other)
Responsible Party: Principal Investigator, Meseret Firde, Prevalence and associated factors of anesthetic drug administration error among anesthetists working in teaching and referral hospitals of Ethiopia, a web based crossectional survey, 2022., DebreTabor University
Other Study IDs: DebreTaborU
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Frequency of Anesthetics Drug Administration Error by Anesthetists
Keywords: Anesthetic drug, medication admnistration, medication admnistration, medication admnistration error
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anesthesia professionals: anesthetists working at teaching and referral hospitals of north west Ethiopia
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — since this is a cross sectional observational study any form of intervention was not applicable

SUMMARY:
The operating room (OR) is a demanding and time-constrained setting, in comparison to primary care settings, where perioperative medication administration is more complicated and there is a high risk that the patient will experience a medication error.

Without consulting the pharmacist or seeking assistance from other staff members, anesthesia clinicians prepare, deliver, and monitor strong anesthetic drugs.

DETAILED DESCRIPTION:
The operating room (OR) is a demanding and time-constrained setting, in comparison to primary care settings, where perioperative medication administration is more complicated and there is a high risk that the patient will experience a medication error. Anesthesia clinicians prepare, deliver, and monitor strong anesthetic drugs without consulting pharmacists or seeking assistance from other staff members.

The aim of this study was to determine the prevalence of medication administration errors by anesthetists and associated factors in referral and teaching hospitals in the Amhara region of, Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* all anesthetists with a minimum of six months of working experience, the ability to respond to the questionnaire using the listed online choices, and involvement in direct patient care to be included in the study.

Exclusion Criteria:

* Anesthetists who were not involved in medication administration and those serving in administrative positions were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all volunteer anesthetists with a minimum of six months of working experience and able to respond to the questionnaire using the listed online choices.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of anesthetics drug administration error by anesthetists working in Amhara region, Ethiopia | October 1-November 30, 2022
  This study aimed to determine the type, frequency, and factors that lead to medication errors in patients under anesthesia.
  This study aimed to determine the type, frequency, and factors that lead to medication errors in patients under anesthesia.
  This study aimed to determine the type, frequency, and factors that lead to medication errors in patients under anesthesia

SECONDARY OUTCOMES:
factors associated with medication administration errors by anesthetists | October 1-November 30, 2022
  This study aimed to determine the type, frequency, and factors that lead to medication errors in patients under anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Debre Tabor University, Debre Tabor, Ethiopia

IPD SHARING:
Plan to Share IPD: No